CLINICAL TRIAL: NCT00259987
Title: A Phase II, Open-Label Study Evaluating Clinical Efficacy, Safety, Pharmacokinetic and Pharmacodynamic Effects of Lapatinib (GW572016) in Patients With Relapsed Adenocarcinoma of the Esophagus, Including Tumors of the Gastroesophageal Junction and Gastric Cardia
Brief Title: Effects Of Lapatinib (GW572016) In Patients With Relapsed Adenocarcinoma Of The Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF102980; NCT00345995 (obsolete NCT alias)
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Adenocarcinoma
Keywords: relapsed adenocarcinoma; esophagus; tumors; GE junction; cancer; lapatinib; gastric cardia
MeSH Terms: conditions — Adenocarcinoma; Neoplasms | interventions — Lapatinib

INTERVENTIONS:
Drug: Lapatinib (GW572016) oral tablets

SUMMARY:
This Phase II study will assess the efficacy, safety, and pharmacodynamics and pharmacokinetics of 1000 mg and 1500 mg lapatinib administered once daily in patients with relapsed adenocarcinoma of the esophagus, including tumors of the GE junction and gastric cardia.

ELIGIBILITY:
Inclusion criteria:

* Has a histologically confirmed adenocarcinoma of the esophagus.
* GE (gastroesophageal) junction or gastric cardia.
* Must be of non-child-bearing potential or is of child-bearing potential.
* Have a negative serum pregnancy test and agree to an approved form of birth control.
* Have an ECOG (Eastern Cooperative Oncology Group) Performance status less than or equal to 2.
* Have a life expectancy of at least 12 weeks.
* Have provided written informed consent.
* Investigator considers patient to be fit for study from lab test results and interview.

Exclusion criteria:

* Pregnant or lactating female.
* Prior resection of the small bowel.
* Received major surgery.
* Received prior radiation therapy to the mediastinum or abdomen.
* Has a known immediate or delayed hypersensitivity reaction.
* Idiosyncrasy to drugs chemically related to the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-11; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) of treatment with daily lapatinib at two different doses (1000 mg and 1500 mg per day) | daily throughout the study

SECONDARY OUTCOMES:
Safety and clinical benefit of lapatinib therapy, progression-free survival, and response duration in the two dose levels combined as well as for the two doses separately. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (6):
- United States (3):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Buffalo, New York
- GSK Investigational Site, Amsterdam, Netherlands
- Peru (2):
  - GSK Investigational Site, San Isidro, Lima region
  - GSK Investigational Site, Lima